CLINICAL TRIAL: NCT01281540
Title: Double-Blind, Randomized, Placebo-Controlled Trial To Assess Efficacy And Safety Of R051619 (Cisapride 10 mg q.i.d.) Versus Placebo For The Improvement Of Symptoms Associated With Exacerbations Of Idiopathic Gastroparesis, After Failure Of Other Treatment Options
Brief Title: An Efficacy and Safety Study of Cisapride in Patients With Chronic Gastroparesis After Failure of Other Treatment Options
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Portfolio/CDT Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR003949; CIS-INT-26
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastroparesis
Keywords: Cisapride ( PREPULSID ); Placebo; Idiopathic; Stomach Diseases; Stomach
MeSH Terms: conditions — Gastroparesis; Stomach Diseases | interventions — Cisapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Cisapride one 10 mg tablet 4 times a day for 8 weeks
  Interventions: Drug: Cisapride
- 002 (Placebo Comparator): Placebo one placebo tablet 4 times a day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cisapride — one 10 mg tablet 4 times a day for 8 weeks
  Arms: 001
Drug: Placebo — one placebo tablet 4 times a day for 8 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to assess the effectiveness of cisapride in patients with a primary diagnosis of chronic gastroparesis (a stomach disorder) of unknown cause.

DETAILED DESCRIPTION:
This is a double-blind (neither the physician nor the patient will know the name of assigned treatment) study to determine the effectiveness of cisapride tablets compared to placebo tablets (a tablet identical in appearance to cisapride but does not contain active drug) in patients with a primary diagnosis of idiopathic gastroparesis (a disorder of unknown cause in which the stomach empties its contents very slowly into the small intestine for digestion. Symptoms of gastroparesis may include vomiting, nausea, early feeling of fullness after only a few bites of food, weight loss due to poor absorption of nutrients or low calorie intake, abdominal bloating, poor glycemic (blood sugar) control, lack of appetite, and pain in the stomach area. Patients will take study drug (one 10-mg tablet of cisapride, or one tablet of placebo), orally, 4 times a day, for a period of 8 weeks. Study drug will be taken approximately 15 minutes before each meal, and, with a beverage, before going to bed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with nondiabetic idiopathic gastroparesis and having symptoms for at least 12 weeks in the preceeding 12 months
* Experienced inadequate response, or intolerance to therapy to date
* Have exacerbation of gastroparesis symptoms requiring medical attention
* Demonstrate delayed gastric emptying as assessed by a [1-13C]-Sodium Acetate Breath Test within 14 days before randomization

Exclusion Criteria:

* Received prior treatment with cisapride
* Have a gycosylated hemoglobin (HbA1c) >7% and bloodglucose of 126 mg/dL (7.0 mmol/L) or greater at screening, as determined by clinical laboratory testing
* Have any upper gastrointestinal (GI) pathology other than idiopathic gastroparesis that would require therapy other than that provided in this trial
* Have any organic/neurological disease that is suspected to be causing gastroparesis
* Currently vomiting, or receiving therapy for a severe exacerbation of gastroparesis, that would prevent the patient from receiving oral therapy or a diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-05; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The average change from baseline in Gastroparesis Cardinal Symptoms Index (GCSI) score | At baseline (Week 0) up to 8 weeks

SECONDARY OUTCOMES:
The number and type of adverse events reported | From time of first dose to the last dose (up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.